CLINICAL TRIAL: NCT03809130
Title: Effectiveness of a Newly Developed Online Intervention on Alleviating Cancer-Related Fatigue in Patients and Survivors
Brief Title: Effectiveness of an Online Intervention Targeting Cancer-related Fatigue
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated Per PI
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0175; NCI-2018-02992 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0175 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Cancer Survivor; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Untire application) (Experimental): Patients use Untire application intervention after baseline up to 6 months.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (Untire application) (Active Comparator): Patients use Untire application intervention after 3 months up to 6 months.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Use Untire application after baseline up to 6 months
  Arms: Arm I (Untire application)
Other: Internet-Based Intervention — Use Untire application after 3 months up to 6 months
  Arms: Arm II (Untire application)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well Untire application intervention works in reducing cancer-related fatigue in cancer patients and survivors.The Untire application focuses on themes that have been identified as causing or contributing to cancer-related fatigue. It may provide information and tips to improve lifestyle, give exercises for body and mind to increase energy levels, offer weekly reports to measure progress, and offer access to an online support community.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the effectiveness of an online multidisciplinary psychological training program delivered via a smartphone-based application (the Untire app) in reducing patient-reported fatigue in cancer patients and survivors.

SECONDARY OBJECTIVES:

I. To determine the dose-response association between use of the Untire app and reduction in patient-reported fatigue severity.

II. To explore whether changes in positive and negative affect, depressive symptoms interact with the effects of the Untire app on fatigue severity.

III. To explore the predictive value of genetic markers (single-nucleotide polymorphisms) and personality characteristics for effectiveness of the Untire app in reducing patient-reported fatigue.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients use Untire application intervention after baseline up to 6 months.

ARM II: Patients use Untire application intervention after 3 months up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present at the Cancer-Related Fatigue Clinic or the Psychiatric Oncology Clinic for an initial consult
* Patients who speak and read English
* Patients who are willing and able to review, understand, and provide written consent
* Patients who agree to comply with all study procedures
* Patients who are in possession of a smartphone or tablet that supports the Untire app software
* Patients rating their current fatigue severity as moderate to severe (= or > 4 on a 0-10 scale), assessed as part of the clinics' screening procedure

Exclusion Criteria:

* Case report of diagnosis of a formal thought disorder (e.g., schizophrenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported fatigue severity as assessed with the Checklist Individual Strength (CIS) between T0 and T1 | Baseline up to 3 months
  The effect of the intervention on fatigue will be analyzed with a generalized linear model, including CIS-20 sum score at T1 as the dependent variable, CIS-20 sum score at T0 as covariate, and group (intervention versus wait-list control) as independent variable.

SECONDARY OUTCOMES:
Total days on which the patient logged in to the app | Up to 6 months
  Change in fatigue between T0 and T1 for the intervention group and between T1 and T2 for the wait-list control group will be entered as dependent variable in multiple regression models, with group allocation as covariate. Separate models will be computed including the different app-usage metrics assessed between T0 -T1 for the intervention group and T1-T2 for the control group as independent variable. These models will additionally be calculated for change in fatigue and use of the app between T0 and T2, for patients in the intervention arm only.
Total number of activities completed on the app | Up to 6 months
  Change in fatigue between T0 and T1 for the intervention group and between T1 and T2 for the wait-list control group will be entered as dependent variable in multiple regression models, with group allocation as covariate. Separate models will be computed including the different app-usage metrics assessed between T0 -T1 for the intervention group and T1-T2 for the control group as independent variable. These models will additionally be calculated for change in fatigue and use of the app between T0 and T2, for patients in the intervention arm only.
Total number of completed assessments on the app | Up to 6 months
  Change in fatigue between T0 and T1 for the intervention group and between T1 and T2 for the wait-list control group will be entered as dependent variable in multiple regression models, with group allocation as covariate. Separate models will be computed including the different app-usage metrics assessed between T0 -T1 for the intervention group and T1-T2 for the control group as independent variable. These models will additionally be calculated for change in fatigue and use of the app between T0 and T2, for patients in the intervention arm only.
Change in negative affect (delta-NA) between T0-T1 | Baseline up to 3 months
  The linear model described for the primary objective will be repeated.
Change in positive affect (delta (PA) between T0-T1 | Baseline up to 3 months
  The linear model described for the primary objective will be repeated.
Change in depressive symptoms (delta-depr) between T0 and T1 | Baseline up to 3 months
  The linear model described for the primary objective will be repeated.
Personality traits | Up to 6 months
  Personality traits and their interaction with group will be added as independent variables to the linear model described for the primary objective.
Genotypes | Up to 6 months
  Genotypes will be dichotomized (presence of minority alleles in the gene of interest) and added as covariates and in interaction with group to the models.

CONTACTS AND LOCATIONS:
Overall Officials: Cobi J Heijnen, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org